| 1 | Design of the pilot, proof of concept REMOTE-COVID trial: |
|---|---|
| 2 | REmote MOniToring usE in suspected cases of COVID-19 |
| 3 | (SARS-CoV 2) |
| 4 | A trial protocol |
| 5 | |
| 6 | Fahad Mujtaba Iqbal <sup>1*</sup> , Meera Joshi <sup>1</sup> , Gary Davies <sup>2</sup> , Sadia Khan <sup>2</sup> , Hutan Ashrafian <sup>1</sup> , Ara Darzi <sup>1</sup> |
| 7<br>8<br>9 | <ol> <li>Division of Surgery &amp; Cancer, 10<sup>th</sup> Floor Queen Elizabeth the Queen Mother Wing (QEQM) St<br/>Mary's Campus, London, W2 1NY</li> <li>West Middlesex University Hospital, Twickenham Road, Isleworth, TW7 6AF</li> </ol> |
| 10 | |
| 11 | |
| 12 | Clinical trials registration information: ClinicalTrials.gov Identifier: NCT04337489 |
| 13 | |
| 14 | 16 March 2020 |
| 15 | |

- 16 Abstract:
- 17 Background: The outbreak of SARS-CoV-2 (coronavirus, COVID-19), declared a pandemic by the
- 18 World Health Organisation (WHO) is global health problem with ever-increasing attributed deaths.
- 19 Vital sign trends are routinely used to monitor patients with changes in these parameters often
- 20 preceding an adverse event. Wearable sensors can measure vital signs continuously (e.g. heart rate,
- 21 respiratory rate, temperature) remotely and can be utilised to recognise early clinical deterioration.
- 22 Methods: We describe the protocol for a pilot, proof-of-concept, observational study to be
- conducted in an engineered hotel near London airports, United Kingdom. The study is set to
- 24 continue for the duration of the pandemic. Individuals arriving to London with mild symptoms
- 25 suggestive of COVID-19 or returning from high risk areas requiring quarantine, as recommended by
- 26 Public Health England, or healthcare professionals with symptoms suggestive of COVID-19 unable to
- isolate at home will be eligible for a wearable patch to be applied for the duration of their stay.
- Notifications will be generated should deterioration be detected through the sensor and displayed
- on a central monitoring hub viewed by nursing staff, allowing for trend deterioration to be noted.
- 30 The primary objective is to determine the feasibility of remote monitoring systems in detecting
- 31 clinical deterioration for quarantined individuals in a hotel.
- 32 Discussion: This trial should prove the feasibility of a rapidly implemented model of healthcare
- delivery through remote monitoring during a global pandemic at a hotel, acting as an extension to a
- 34 healthcare trust. Potential benefits would include reducing infection risk of COVID-19 to healthcare
- 35 staff, with earlier recognition of clinical deterioration through ambulatory, continuous, remote
- 36 monitoring using a discrete wearable sensor. We hope our results can power future, robust future
- 37 randomised trials.
- 38 Trial registration: ClinicalTrials.gov Identifier: NCT04337489
- 39 Keywords: remote sensing technology; protocol; clinical trial; patient deterioration; monitoring,
- 40 ambulatory.

- 41 Background:
- 42 The recent outbreak of SARS-CoV-2 (COVID-19), declared a pandemic by the World Health
- 43 Organisation (WHO) and a growing global health problem, has stretched resources, creating
- 44 pressures within the National Health Service (NHS) with implications for patient safety. 1 UK Chief
- 45 Medical Officers have raised the risk to the UK to high, with ever increasing confirmed cases and
- 46 attributed deaths.<sup>1</sup>
- 47 High risk travellers with suspected or confirmed cases of COVID-19 are likely to transferred
- immediately to hospital. However, travellers with milder symptoms or returning from high risk
- 49 areas, a two-week period of observation/quarantine may be required, in accordance with Public
- 50 Health England recommendations.<sup>2</sup> The rate of clinical deterioration for individuals suffering with
- 51 COVID-19 remains unknown; given that widespread vaccine deployment remains imminently
- 52 unforeseeable, novel strategies are required in approaching this pandemic.
- 53 Vital signs trends (heart rate, respiratory rate, blood pressure, temperature, oxygen saturations) are
- routinely used for monitoring hospital patients.<sup>3</sup> Clinical deterioration may be recognised through
- changes in these parameters, and often precedes an adverse event.<sup>4,5</sup> As such, The National
- Institute for Health and Care Excellence (NICE) and the Royal College of Physicians (RCP) recommend
- that all patients have their vital signs recorded every 12h as a minimum.<sup>6,7</sup>
- Across the National Health Service (NHS), the use of the National Early Warning Score 2 (NEWS), a
- 59 'track and trigger' warning score, has been implemented in accordance with the RCP to guide on
- escalation protocols and monitoring frequency of vital signs. Accordingly, heart rate (HR),
- 61 respiratory rate (RR), temperature, blood pressure, oxygen saturations, and level of consciousness
- are assessed every 4-6 hours with more frequent monitoring for acutely unwell patients.
- Progression in non-invasive digital technologies have renewed potential for remote monitoring
- 64 solutions.<sup>8,9</sup> Wearable sensors offer an opportunity for sensor alerting systems to continuously
- 65 monitor vital parameters remotely, recognise early deterioration and support clinical decision

66 making, allowing people to receive monitoring outside of expensive hospital facilities; in resource

67 limited hospitals; and utilising alternate sites in crisis scenarios. 10

Previous studies have demonstrated acceptability and practicability of continuous monitoring using

wearable sensors on general surgical and medical wards in the UK and The Netherlands. 11,12 Initial

work by Downey et al. were limited by imbalanced randomisation leading to significant baseline

differences across the two trial arms and failure to adjust for these in their analyses. 11 Nevertheless,

the wearable sensor seemed to demonstrate feasibility in hospital settings. Qualitative analyses,

through semi-structured interviews for patients and healthcare staff, similarly favoured continuous

the notion of continuous vital sign monitoring in general wards. 12 It should be noted that many of

the patients interviewed were admitted for malignant disease which is likely to influence qualitative

outcomes. Delivery of healthcare outside of hospital facilities (e.g. in hotels) is theoretically possible

through continuous remote monitoring of vital signs but has yet to be studied; given the global

pandemic and fear of future waves, evaluation of its viability is justified.

79 Here, we describe the design of our pragmatic trial, exploring the feasibility of remote monitoring

systems in suspected cases of COVID-19 at a hotel, primarily as earlier recognition of clinical

deterioration.

68

69

70

71

72

73

74

75

76

77

78

80

81

- Methods:
- 83 Overall design:
- 84 This pragmatically designed, pilot, proof-of-concept, observational study was reviewed and
- 85 approved by London Queen Square Research Ethics Committee (IRAS: 281757) and this protocol
- 86 was developed in accordance with recommendations from the Standard Protocol Items:
- 87 Recommendations for Interventional Trials (SPIRIT) guidelines.<sup>13</sup> The objective is to determine the
- feasibility of remote healthcare delivery in a hotel with rapid implementation in the COVID-19 era.
- 89 Feasibility will be tested through rate of participation and number of vital alerts generated.

The SensiumVitals™ (Sensium Healthcare Ltd., United Kingdom) system can be engineered in the building (hotel) for use with the wearable sensor. All participants would be fitted with the sensor on arrival and would always be worn. A designated area within the facility would act as a central hub allowing for remote monitoring to occur by healthcare staff. Alerts would be generated, in accordance with NEWS parameters (Table 1) but can be individually tailored, to identify deteriorating participants. Participants can be escalated to hospitals should rapid deteriorating in vital signs be noted; ambulance services and paramedics will be present on site to facilitate this. The decision to escalate will come from a senior nurse, present on site, or a general practitioner contactable at all times.. The temperature alert threshold was lowered to the lowest score in the NEWS chart, allowing for earlier detection and improved sensitivity¹⁴; this decision was made from previous work which demonstrated varying limits of agreement for temperature when compared to nursing observations.¹¹⁵ Escalation protocols will be developed and trialled, allowing staff to address issues as they arise (Figure 1).

Wearable sensor system

SensiumVitals™ by the Surgical Company, have produced a lightweight, waterproof, single-use, wearable wireless 'patch' with a battery life of 5 days measuring vital signs every two minutes. The sensor attaches to an individual's chest with two ECG electrodes, recording HR, RR, and a wire attaches around the individual's back, measuring axillary temperature. The sensor is FDA approved and CE marked. Data are transmitted through radiofrequency and dedicated intranet hotspots. Physiological parameters can be viewed by clinical staff on a mobile device/desktop computer, allowing trends towards deterioration to be noted, with tailored alerts generated for deteriorating individuals in accordance with NEWS (Figure 2).

All sensor data collected by the SensiumVitals® system will be stored on a created secured hotel network; access to which is restricted to research personnel. Given that the hotel acts as an

extension to a healthcare trust, the SensiumVitals® system inherits all the hospital procedures and data backup policies, ensuring data access and servers are secured.

In line with the principles of Good Clinical Practice guidelines, data will be securely archived for a minimum of 5 years.

Following the completion of quarantine, participants will be invited to share their experiences through using semi-structured interviews and questionnaires. Individual interviews allow for anonymity and truthful perceptions/attitudes. This method enables narratives to be elicited through guided but open questioning.

### Hypotheses:

116

117

118

119

120

121

122

123

124

125

126

128

129

130

131

132

133

134

135

136

137

- Continuous remote monitoring with wearable sensors of vital signs will identify deteriorating patients.
- Healthcare provision in a hotel will be feasible and acceptable amongst healthcare staff and participants.

### **127** *Sequence of events:*

# Patching patients and using data for academic research

- 1. Eligible participants from the airport will be transferred to the hotel by paramedics.
- Upon arrival to the engineered hotel, an initial assessment of all participants will be undertaken. A study information sheet will be provided, and informed consent taken for wearable sensors to be applied, allowing remote monitoring of vital signs. To ensure appropriate quarantine.
  - 3. In a designated area within the building, a central monitoring hub will be set up to monitor the recorded parameters by National Health Service (NHS) healthcare staff from a local Trust. The hub contains a site manager, porters, security staff, nurses, ambulance services, professional cleaners, and hotel staff.

- 4. If a participant deteriorates, an alert should be generated on a smartphone device/desktop computer; following this, an escalation protocol will be trialled to action the alert in an appropriate manner; hospitalisation may be necessary. Initially, nursing staff will gather more information through telephone review. Following this, a virtual GP can be contacted for further advice. Ambulance services and paramedics will be on-site to facilitate hospitalisation should rapid deterioration occur. These healthcare professionals are independent and can provide oversight.
  - 5. Participants will be invited for an interview and be asked to complete a survey on their experiences following quarantine completion.
  - 6. Participant care records will be stored on an online Care Information Exchange system (compliant with General Data Protection Regulation) that is currently in place across the trust. Electronic health records and patient notes will be reviewed to determine clinically relevant events if transfer to hospital occurs (e.g. hospital length of stay, mortality, escalation to ITU).
  - 7. Sensor data will be extracted from the central servers containing sensor data for appropriate statistical analyses for associated clinical efficacy of health outcomes in COVID-19.

## <u>Semi-structured interviews/Questionnaires (mixed methods)</u>

- All participants alongside healthcare staff will be invited to take part in semi-structured interviews and be given questionnaires. These will take place by the primary lead researcher using prepared topic guides.
- 2. Written consent will be obtained from those who agree to participate.
- 3. An audio recording will be made of the interviews. Notes reflecting verbal responses may be
   taken. The interviews will be conducted at the engineered hotel.
  - 4. The recordings will be transcribed, and the data will undergo thematic analyses.

145

146

147

148

149

150

151

152

153

154

155

156

157

158

159

| 163 | 5. | Validated and unvalidated questionnaires will also be given enquiring about experiences |
|---|---|---|
| 164 | | (e.g. PHQ-9 <sup>16</sup> , GAD-7 <sup>17</sup> , satisfaction, anxiety related to the devices). |
| 165 | | |
| 166 | Outcor | nes and progression criteria: |
| 167 | <u>Feasibil</u> | ity outcomes: |
| 168 | 1. | Rate of participation |
| 169<br>170 | | Using the confidence interval approach <sup>18</sup> , for a minimum sample size of 10 individuals, we estimate a rate of participation of 90% with a 95% confidence interval of +/- 18%. |
| 171<br>172 | 2. | Generation of an alert following abnormal vital signs (e.g. raised temperature). We aim for a minimum of 5 vital alerts to be generated to demonstrate feasibility. |
| 173<br>174 | 3. | Missing data recorded from sensor limited to less than 20% attrition will be a criterion for progression. |
| 175 | 4. | Number of adverse events relating to the sensor system (e.g., skin reaction to sensor |
| 176 | | preventing trial continuation) |
| 177 | | |
| 178 | Explora | tory clinical outcomes: |
| 179 | 1. | Actions following alert generation (e.g., phone consultation, virtual general practitioner |
| 180<br>181 | 2. | review, transfer to hospital). Acceptability and usability of the SensiumVitals™ system by healthcare staff and participants |
| 182 | | (mixed methods analysis) |
| 183 | | |
| 184 | Partici | pant eligibility: |
| 185 | The stu | dy will recruit flight arrivals returning to the UK in London. High risk travellers are screened |
| 186 | at the airport and tested for COVID-19, with transfer to hospital if appropriate; this cohort would be | |
| 187 | ineligib | le for the study. |
| 188 | Additio | nally, healthcare professionals who display symptoms of COVID-19 and are unable to isolate |
| 189 | safely a | t home (e.g. lodging with vulnerable persons) would be eligible to take part in the study and |
| 190 | invited | to stay at the hotel. |
| 191 | Inclusio | on Criteria |

192

• Aged 18 years or over.

- Able to provide written consent.
- Travellers returning with milder symptoms suggestive of COVID-19 or returning from high
   risk areas requiring quarantine, as recommended by Public Health England.
  - Healthcare professionals with milder symptoms suggestive of COVID-19 unable to isolate at home.

#### **Exclusion Criteria**

196

197

198

203

204

205

206

208

209

210

211

212

213

214

215

216

- Any participants that withdraw their consent.
- A skin condition/reaction preventing wearing the wearable sensor (these can be communicated by the participant to the researcher or healthcare staff at the hotel).
- The presence of a permanent pacemaker or cardiac defibrillator.
  - Any form of psychiatric disorder or a condition that, in the opinion of the investigator, may hinder communication with the research team.
    - Inability to cooperate or communicate with the research team.

207 Statistical considerations:

#### Quantitative analysis:

Descriptive statistics will be obtained about the baseline characteristics of participants. Continuous variables will be presented as mean ± standard deviation or medians and ranges, depending on distribution. Categorical variables will be reported as numbers and percentages. The total frequencies of alerts, proportion of actioned alerts, and resultant actions will be described.

Outcome measures (e.g. phone consultation, virtual GP review, transfer to hospital) will be reviewed from case notes should escalation occur and described in absolute frequencies. Questionnaire data will be presented using frequency distributions. Data will be analysed using SPSS, Stata, and GraphPad.

## Qualitative analyses:

Semi structured interviews will take place by the primary lead researcher using the prepared topic guides. An audio recording will be made of all interviews. The interviewer may also take field notes reflecting the verbal responses and reflections to be used to adapt the topic/study direction. The audio recordings will be transcribed. The data will be analysed appropriately using thematic analysis.

To ensure confidentiality and anonymity, each interview will be allocated a pseudonym, to be applied to the corresponding consent form, topic guide form/field notes and audio file. Their name will not be included in the audio recording; the pseudonym will be used.

Summaries of interview field notes will be typed into a word processor. All paper and soft copies of field notes, audio files and consent forms will be kept securely in a locker within a locked office and if in digital format, on a password protected computer and backed up regularly. Information will only be shared within the study team.

Audio recordings will be professionally transcribed verbatim, and a random selection of transcripts will be checked against recordings for accuracy. Interview transcripts will be analysed using Braun and Clarke's thematic analysis by two independent researchers; disagreements will be resolved through discussion.<sup>19</sup> Power considerations:

As a pilot study in an unknown viral pandemic, the progression of which is not well established, this study will appraise the feasibility for hotel remote sensing under these circumstances. Sufficient other data do not exist to allow for power calculations.

### Patient and public involvement:

Due to the nature of the pandemic and the current climate (national lockdown advised from the government) with COVID-19, patient and public involvement was not undertaken for this

observational trial. All eligible participants will be approached to enter the study and all recruited participants can provide email addresses should they wish for dissemination of results.

# Discussion:

240

241

242

243

244

245

246

247

248

249

250

251

252

253

254

255

256

257

258

259

260

261

262

263

264

To the best of our knowledge, this is the first remote monitoring study focussing on healthcare delivery during a global pandemic at a remote site (i.e. hotel), acting as an extension to a healthcare trust. Apart from reducing infection risk to healthcare staff, continuous remote monitoring using a discrete wearable sensor has the potential to detect earlier clinical deterioration allowing for earlier intervention and provide further insight into the clinical course of COVID-19 in regards to vital signs. Our pilot study design will test the viability of using a remote site for healthcare delivery during times of crisis. Continuous vital sign monitoring should provide insight to determine whether vital sign trends can detect clinical deterioration for COVID-19, requiring hospitalisation. Furthermore, questionnaires and semi-structured interviews of participants will provide insight into wider implementation of this technology and provide feedback for improvements. Similarly, semistructured interviews of staff will provide a healthcare perspective, particularly thoughts on reducing potential infection risk through remote monitoring services. Despite the strengths of our study, the design presents inherent limitations. Mainly, the lack of randomisation and control arm to compare remote monitoring services to 'standard care'. However, to maximise capacity at the hotel given the unknown of the pandemic, a pragmatic, observational design was favoured; randomisation was not deemed appropriate. Government restrictions are rapidly changing for air travel, which could significantly alter our sample size, increasing the risk of type II errors. The inclusion of healthcare professionals may bias the description of favourable experiences, owing to their familiarity of continuous monitoring of physiological parameters. In addition, implementing remote monitoring systems entails an initial financial cost with new logistical and legal considerations; given the early phase of work, the true

extent of these issues remains unknown. If the trial is proven to be feasible, this work could power

| 265 | future randomised trials to explore for cause-effect relationships and describe cost- |
|---|---|
| 266 | utility/effectiveness of remote monitoring solutions. |
| 267 | In conclusion, the results of our study would have potential to demonstrate the feasibility of remote |
| 268 | monitoring during a pandemic and may provide insight into earlier recognition of clinical |
| 269 | deterioration in individuals suspected with COVID-19. |
| 270 | |

- 271 Declarations
- 272 Ethics approval and consent to participate
- 273 All participants must provide consent to participate. This study has been received ethical approval
- by London Queen Square Research Ethics Committee (IRAS: 281757).
- **275** *Consent for publication*
- 276 Consent will be taken for publication.
- **277** Availability of data and materials
- The datasets used and/or analysed during the current study are available from the corresponding
- author on reasonable request. Only the authors have access to the dataset.
- **280** *Competing interests*
- 281 The authors declare that they have no competing interests
- 282 Funding
- 283 This work was supported by a grant provided through CW+ (the official charity of Chelsea and
- Westminster Hospital). The funding body will play no role in the design of the study and collection,
- analysis, and interpretation of data and in writing this manuscript.
- 286 Authors' contributions
- 287 FMI drafted the manuscript. Amendments were made by MJ, SK, HA, GD, and AD. Statistical
- considerations were discussed with MJ, SK and HA. The idea was conceived by MJ and SK.
- 289 Acknowledgements
- 290 Infrastructure support for this research was provided by the NIHR Imperial Biomedical Research
- 291 Centre (BRC) and the NIHR Imperial Patient Safety Translational Research Centre (PSTRC).

# 293 References:

- Department of Health and Social Care; Public Health England. Coronavirus (COVID-19): latest
   information and advice GOV.UK. https://www.gov.uk/guidance/coronavirus-covid-19 information-for-the-public. Accessed March 6, 2020.
- 297 2. Public Health England. Stay at home: guidance for households with possible coronavirus
  298 (COVID-19) infection GOV.UK. https://www.gov.uk/government/publications/covid-19-stay299 at-home-guidance/stay-at-home-guidance-for-households-with-possible-coronavirus-covid300 19-infection. Published 2020. Accessed May 6, 2020.
- 301 3. Kenzaka T, Okayama M, Kuroki S, et al. Importance of vital signs to the early diagnosis and severity of sepsis: association between vital signs and sequential organ failure assessment score in patients with sepsis. *Intern Med.* 2012;51(8):871-876.
- Smith GB. In-hospital cardiac arrest: is it time for an in-hospital 'chain of prevention'?
   *Resuscitation*. 2010;81(9):1209-1211.
- DeVita MA, Smith GB, Adam SK, et al. "Identifying the hospitalised patient in crisis"—a
   consensus conference on the afferent limb of rapid response systems. *Resuscitation*.
   2010;81(4):375-382.
- 309 6. National Institutes of Clinical Excellence. Acutely Ill Patients in Hospital: Recognition of and

| 311<br>312<br>313 | 7. | Royal College of Physicians. National Early Warning Score (NEWS) 2. https://www.rcplondon.ac.uk/projects/outputs/national-early-warning-score-news-2. Published 2017. Accessed March 6, 2020. |
|---|---|---|
| 314<br>315<br>316 | 8. | Bombaci A, Abbadessa G, Trojsi F, Leocani L, Bonavita S, Lavorgna L. Telemedicine for management of patients with amyotrophic lateral sclerosis through COVID-19 tail. <i>Neurol Sci.</i> 2020. doi:10.1007/s10072-020-04783-x |
| 317<br>318 | 9. | De Farias FACD, Dagostini CM, Bicca YDA, Falavigna VF, Falavigna A. Remote patient monitoring: A systematic review. <i>Telemed e-Health</i> . 2020. doi:10.1089/tmj.2019.0066 |
| 319<br>320 | 10. | Martirosyan M, Caliskan K, Theuns DAMJ, Szili-Torok T. Remote monitoring of heart failure: benefits for therapeutic decision making. <i>Expert Rev Cardiovasc Ther</i> . 2017;15(7):503-515. |
| 321<br>322<br>323 | 11. | Downey C, Randell R, Brown; Julia, Jayne DG. Continuous Versus Intermittent Vital Signs Monitoring Using a Wearable, Wireless Patch in Patients Admitted to Surgical Wards: Pilot Cluster Randomized Controlled Trial. <i>J Med Internet Res.</i> 2018;20(12). doi:10.2196/10802 |
| 324<br>325<br>326 | 12. | Weenk M, Bredie SJ, Koeneman M, Hesselink G, van Goor H, van de Belt TH. Continuous Monitoring of Vital Signs in the General Ward Using Wearable Devices: Randomized Controlled Trial. <i>J Med Internet Res</i> . 2020;22(6):e15471. doi:10.2196/15471 |
| 327<br>328<br>329 | 13. | Chan A-W, Tetzlaff JM, Altman DG, et al. SPIRIT 2013 Statement: Defining Standard Protocol Items for Clinical Trials. <i>Ann Intern Med.</i> 2013;158(3):200-207. doi:10.7326/0003-4819-158-3 201302050-00583 |
| 330<br>331 | 14. | Royal College of Physicians. National Early Warning Score (NEWS) 2 RCP London. <i>NEWS 2</i> . 2017. |
| 332<br>333<br>334<br>335 | 15. | Downey C, Ng S, Jayne D, Wong D. Reliability of a wearable wireless patch for continuous remote monitoring of vital signs in patients recovering from major surgery: a clinical validation study from the TRaCINg trial. <i>BMJ Open</i> . 2019;9(8):e031150. doi:10.1136/bmjopen-2019-031150 |
| 336<br>337 | 16. | Kroenke K, Spitzer RL, Williams JBW. The PHQ-9: validity of a brief depression severity measure. <i>J Gen Intern Med</i> . 2001;16(9):606-613. |
| 338<br>339<br>340 | 17. | Spitzer RL, Kroenke K, Williams JBW, Löwe B. A Brief Measure for Assessing Generalized Anxiety Disorder: The GAD-7. <i>Arch Intern Med</i> . 2006;166(10):1092-1097. doi:10.1001/archinte.166.10.1092 |
| 341<br>342 | 18. | Thabane L, Ma J, Chu R, et al. A tutorial on pilot studies: the what, why and how. <i>BMC Med Res Methodol</i> . 2010;10(1):1. doi:10.1186/1471-2288-10-1 |
| 343<br>344 | 19. | Braun V, Clarke V. Using thematic analysis in psychology. <i>Qual Res Psychol</i> . 2006;3(2):77-101. doi:10.1191/1478088706qp063oa |
| 345 | | |
| 346<br>347 | Figure legends: Figure 1: Potential escalation pathway; NEWS: National Early Warning Score; GP: general | |
| 348 | practi | tioner. |

Response to Acute Illness in Adults in Hospital. National Institute for Clinical Excellence; 2007.

Figure 2: Monitoring system for SensiumVitals™ Wearable Sensor

350 Table:

351

Table 1: Criteria for generating vitals alert

| Parameter | Alert threshold |
|---------------------------------------|-----------------|
| Respiratory rate (breaths per minute) | <u>&gt;</u> 25 |
| Temperature (Celsius) | <u>≥</u> 38.1 |
| Heart rate (beats per minute) | <u>&gt;</u> 131 |

352